CLINICAL TRIAL: NCT04037163
Title: CCTA-FFR Registry for Development of Comprehensive Risk Prediction Model
Brief Title: CCTA-FFR Registry for Risk Prediction
Status: Completed | Type: Observational
Sponsor: Seoul National University Hospital (Other)
Collaborators: Keimyung University Dongsan Medical Center (Other); Inje University (Other); Tsuchiura Kyodo General Hospital (Other)
Responsible Party: Principal Investigator, Bon-Kwon Koo, Professor, Seoul National University Hospital
Other Study IDs: H-1907-094-1048
Record Dates: First submitted 2019-07-22; First posted 2019-07-30 (Actual); Last update posted 2019-07-30 (Actual); Status verified 2019-07

CONDITIONS: Coronary Artery Disease
Keywords: Fractional flow reserve; Coronary CT angiography; Atherosclerosis
MeSH Terms: conditions — Coronary Artery Disease; Atherosclerosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- CCTA-FFR: Patients who underwent CCTA within 90 days before FFR measurement will be included in the present study.
  Interventions: Diagnostic Test: Fractional flow reserve, Coronary CT angiography

INTERVENTIONS:
Diagnostic Test: Fractional flow reserve, Coronary CT angiography — Coronary CT angiography was performed as part of routine clinical practice for patients with suspected coronary artery disease and the decision to perform coronary CT angiography before invasive angiography was at the judgment of the physicians in charge.

SUMMARY:
The investigators sought to investigate the prognostic implication of qualitative and quantitative plaque analysis on coronary CT angiography (CCTA) according to fractional flow reserve (FFR). The main objective was to develop a comprehensive risk model by using clinical risk factors, FFR and CCTA parameters.

DETAILED DESCRIPTION:
Coronary CT angiography (CCTA) is an evolving noninvasive modality in diagnosis of coronary artery disease (CAD). Its incremental prognostic value over traditional scheme of risk prediction has repeatedly been demonstrated. Beyond the assessment of CAD severity, the prognostic value of CCTA has increased with comprehensive plaque analysis. Certain plaque features on CCTA have a prognostic value in the prediction of future coronary events. The concept of fractional flow reserve (FFR) has been developed as an invasive index of the functional severity of stenosis. FFR represents maximal blood flow to the myocardium supplied by an artery with stenosis as a fraction of normal maximum flow. In moderate stenotic lesion, determining whether to perform PCI based on FFR is a current guideline, and has been proven to reduce unnecessary revascularization procedure and improve clinical prognosis. However, clinical events still occur in patients with FFR >0.80. In a recent study, the prognosis in the vessel with FFR > 0.8 was investigated. However, a comprehensive risk model according to FFR has never been investigated. Therefore, the investigators sought to investigate the prognostic implication of qualitative and quantitative plaque analysis on CCTA according to FFR. The main objective was to develop a comprehensive risk model by using clinical risk factors, FFR, and CCTA parameters.

Patients who underwent CCTA within 90 days before FFR measurement will be included. The study population will be from 2 different registries. The 3V-FFR-FRIENDS registry (NCT0620122050) enrolled a total of 1,136 patients (3,298 vessels). Among them, 299 patients who underwent CCTA within 90 days before FFR measurement will be included. The institutional registry of Tsuchiura Kyodo General Hospital included 448 patients who underwent FFR measurement and CCTA within 90 days. By retrospectively collecting clinical outcome data, coronary angiographic data, physiologic indices, and CCTA data from two registries, the CCTA-FFR Registry for Development of Comprehensive Risk Prediction Model will be created. For 3V FFR-FRIENDS registry (NCT0620122050), the collected clinical data for the previous study will be used, and 5-year outcome data will be collected from Seoul National University Hospital, Keimyung University Dongsan Medical Center, and Inje University Ilsan Paik Hospital. For the Institutional registry of Tsuchiura Kyodo General Hospital registry, the investigators will collect the baseline characteristics of participants, CCTA data, and clinical outcome data followed until Mar 2019.

ELIGIBILITY:
Inclusion Criteria:

* Patients who underwent CCTA within 90 days before FFR measurement

Exclusion Criteria:

* Unanalyzable coronary CT angiography
* Inadequate fractional flow reserve measurement

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with suspected coronary artery disease who underwent coronary CT angiography within 90 days before FFR measurement will be included.
Sampling Method: Non-Probability Sample
Enrollment: 747 (Actual)
Dates: Start 2010-12-22 (Actual); Primary Completion 2019-03-31 (Actual); Study Completion 2019-05-31 (Actual)

PRIMARY OUTCOMES:
Discrimination index of prediction model for vessel-oriented composite outcome | Upto 5 years after index procedure
  A risk model for vessel-oriented composite outcome, incorporating clinical, angiographic, fractional flow reserve (FFR), and coronary CT angiographic parameters will be developed. Vessel-oriented composite outcome is a composite of cardiac death, vessel-related myocardial infarction (MI), or vessel-related ischemia-driven revascularization. The target vessel will be defined as the vessel with FFR measurement.

CONTACTS AND LOCATIONS:
Overall Officials: Bon-Kwon Koo, MD, PhD, Study Director — Seoul National University Hospital; Joon Hyung Doh, MD, PhD, Principal Investigator — Inje University; Chang-Wook Nam, MD, PhD, Principal Investigator — Keimyung University Dongsan Medical Center; Tsunekazu Kakuta, MD, PhD, Principal Investigator — Tsuchiura Kyodo General Hospital

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Nielsen LH, Botker HE, Sorensen HT, Schmidt M, Pedersen L, Sand NP, Jensen JM, Steffensen FH, Tilsted HH, Bottcher M, Diederichsen A, Lambrechtsen J, Kristensen LD, Ovrehus KA, Mickley H, Munkholm H, Gotzsche O, Husain M, Knudsen LL, Norgaard BL. Prognostic assessment of stable coronary artery disease as determined by coronary computed tomography angiography: a Danish multicentre cohort study. Eur Heart J. 2017 Feb 7;38(6):413-421. doi: 10.1093/eurheartj/ehw548. PMID 27941018
- [Background] Cho I, Al'Aref SJ, Berger A, O Hartaigh B, Gransar H, Valenti V, Lin FY, Achenbach S, Berman DS, Budoff MJ, Callister TQ, Al-Mallah MH, Cademartiri F, Chinnaiyan K, Chow BJW, DeLago A, Villines TC, Hadamitzky M, Hausleiter J, Leipsic J, Shaw LJ, Kaufmann PA, Feuchtner G, Kim YJ, Maffei E, Raff G, Pontone G, Andreini D, Marques H, Rubinshtein R, Chang HJ, Min JK. Prognostic value of coronary computed tomographic angiography findings in asymptomatic individuals: a 6-year follow-up from the prospective multicentre international CONFIRM study. Eur Heart J. 2018 Mar 14;39(11):934-941. doi: 10.1093/eurheartj/ehx774. PMID 29365193
- [Background] SCOT-HEART Investigators; Newby DE, Adamson PD, Berry C, Boon NA, Dweck MR, Flather M, Forbes J, Hunter A, Lewis S, MacLean S, Mills NL, Norrie J, Roditi G, Shah ASV, Timmis AD, van Beek EJR, Williams MC. Coronary CT Angiography and 5-Year Risk of Myocardial Infarction. N Engl J Med. 2018 Sep 6;379(10):924-933. doi: 10.1056/NEJMoa1805971. Epub 2018 Aug 25. PMID 30145934
- [Background] Motoyama S, Ito H, Sarai M, Kondo T, Kawai H, Nagahara Y, Harigaya H, Kan S, Anno H, Takahashi H, Naruse H, Ishii J, Hecht H, Shaw LJ, Ozaki Y, Narula J. Plaque Characterization by Coronary Computed Tomography Angiography and the Likelihood of Acute Coronary Events in Mid-Term Follow-Up. J Am Coll Cardiol. 2015 Jul 28;66(4):337-46. doi: 10.1016/j.jacc.2015.05.069. PMID 26205589
- [Background] Williams MC, Moss AJ, Dweck M, Adamson PD, Alam S, Hunter A, Shah ASV, Pawade T, Weir-McCall JR, Roditi G, van Beek EJR, Newby DE, Nicol ED. Coronary Artery Plaque Characteristics Associated With Adverse Outcomes in the SCOT-HEART Study. J Am Coll Cardiol. 2019 Jan 29;73(3):291-301. doi: 10.1016/j.jacc.2018.10.066. PMID 30678759
- [Background] De Bruyne B, Baudhuin T, Melin JA, Pijls NH, Sys SU, Bol A, Paulus WJ, Heyndrickx GR, Wijns W. Coronary flow reserve calculated from pressure measurements in humans. Validation with positron emission tomography. Circulation. 1994 Mar;89(3):1013-22. doi: 10.1161/01.cir.89.3.1013. PMID 8124786
- [Background] Berger A, Botman KJ, MacCarthy PA, Wijns W, Bartunek J, Heyndrickx GR, Pijls NH, De Bruyne B. Long-term clinical outcome after fractional flow reserve-guided percutaneous coronary intervention in patients with multivessel disease. J Am Coll Cardiol. 2005 Aug 2;46(3):438-42. doi: 10.1016/j.jacc.2005.04.041. PMID 16053955
- [Background] Tonino PA, De Bruyne B, Pijls NH, Siebert U, Ikeno F, van' t Veer M, Klauss V, Manoharan G, Engstrom T, Oldroyd KG, Ver Lee PN, MacCarthy PA, Fearon WF; FAME Study Investigators. Fractional flow reserve versus angiography for guiding percutaneous coronary intervention. N Engl J Med. 2009 Jan 15;360(3):213-24. doi: 10.1056/NEJMoa0807611. PMID 19144937
- [Background] Pijls NH, van Son JA, Kirkeeide RL, De Bruyne B, Gould KL. Experimental basis of determining maximum coronary, myocardial, and collateral blood flow by pressure measurements for assessing functional stenosis severity before and after percutaneous transluminal coronary angioplasty. Circulation. 1993 Apr;87(4):1354-67. doi: 10.1161/01.cir.87.4.1354. PMID 8462157
- [Background] Park J, Lee JM, Koo BK, Shin ES, Nam CW, Doh JH, Hwang D, Zhang J, Hu X, Wang J, Ye F, Chen S, Yang J, Chen J, Tanaka N, Yokoi H, Matsuo H, Takashima H, Shiono Y, Akasaka T. Clinical Relevance of Functionally Insignificant Moderate Coronary Artery Stenosis Assessed by 3-Vessel Fractional Flow Reserve Measurement. J Am Heart Assoc. 2018 Feb 15;7(4):e008055. doi: 10.1161/JAHA.117.008055. PMID 29449274
- [Derived] Kim CH, Yang S, Zhang J, Lee JM, Hoshino M, Murai T, Hwang D, Shin ES, Doh JH, Nam CW, Wang J, Chen SL, Tanaka N, Matsuo H, Akasaka T, Kakuta T, Koo BK. Differences in Plaque Characteristics and Myocardial Mass: Implications for Physiological Significance. JACC Asia. 2022 Mar 29;2(2):157-167. doi: 10.1016/j.jacasi.2021.11.011. eCollection 2022 Apr. PMID 36339124
- [Derived] Yang S, Lee JM, Hoshino M, Murai T, Choi KH, Hwang D, Kim KJ, Shin ES, Doh JH, Chang HJ, Nam CW, Zhang J, Wang J, Chen SL, Tanaka N, Matsuo H, Akasaka T, Kakuta T, Koo BK. Prognostic Implications of Comprehensive Whole Vessel Plaque Quantification Using Coronary Computed Tomography Angiography. JACC Asia. 2021 Jun 15;1(1):37-48. doi: 10.1016/j.jacasi.2021.05.003. eCollection 2021 Jun. PMID 36338359
- [Derived] Yang S, Hoshino M, Yonetsu T, Zhang J, Hwang D, Shin ES, Doh JH, Nam CW, Wang J, Chen S, Tanaka N, Matsuo H, Kubo T, Chang HJ, Kakuta T, Koo BK. Outcomes of non-ischaemic coronary lesions with high-risk plaque characteristics on coronary CT angiography. EuroIntervention. 2023 Jan 23;18(12):1011-1021. doi: 10.4244/EIJ-D-22-00562. PMID 36222756
- [Derived] Yang S, Hoshino M, Koo BK, Yonetsu T, Zhang J, Hwang D, Shin ES, Doh JH, Nam CW, Wang J, Chen S, Tanaka N, Matsuo H, Kubo T, Chang HJ, Kakuta T, Narula J. Relationship of Plaque Features at Coronary CT to Coronary Hemodynamics and Cardiovascular Events. Radiology. 2022 Dec;305(3):578-587. doi: 10.1148/radiol.213271. Epub 2022 Aug 16. PMID 35972355
- [Derived] Yang S, Koo BK, Hwang D, Zhang J, Hoshino M, Lee JM, Murai T, Park J, Shin ES, Doh JH, Nam CW, Wang J, Chen S, Tanaka N, Matsuo H, Akasaka T, Chang HJ, Kakuta T, Narula J. High-Risk Morphological and Physiological Coronary Disease Attributes as Outcome Markers After Medical Treatment and Revascularization. JACC Cardiovasc Imaging. 2021 Oct;14(10):1977-1989. doi: 10.1016/j.jcmg.2021.04.004. Epub 2021 May 19. PMID 34023270
- [Derived] Yang S, Koo BK, Hoshino M, Lee JM, Murai T, Park J, Zhang J, Hwang D, Shin ES, Doh JH, Nam CW, Wang J, Chen S, Tanaka N, Matsuo H, Akasaka T, Choi G, Petersen K, Chang HJ, Kakuta T, Narula J. CT Angiographic and Plaque Predictors of Functionally Significant Coronary Disease and Outcome Using Machine Learning. JACC Cardiovasc Imaging. 2021 Mar;14(3):629-641. doi: 10.1016/j.jcmg.2020.08.025. Epub 2020 Nov 25. PMID 33248965